CLINICAL TRIAL: NCT05416736
Title: The Effect of Bladder Stimulation Technique on Urine Specimen Collection in Newborns: A Randomized Controlled Study
Brief Title: The Effect of Bladder Stimulation Technique on Urine Specimen Collection in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nihan Korkmaz, Research assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Nihan
Record Dates: First submitted 2022-06-09; First posted 2022-06-13 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Urine Specimen Collection
Keywords: urine specimen; bladder stimulation technique; newborn; comfort; physiological parameters

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): * Newborns will be fed with formula or breast milk pumped, according to the age and weight of the baby.
  * Before the procedure, the newborn's heart rate, saturation and comfort scale score will be recorded.
  * Genital area will be cleaned.
  * Newborn will be held under the armpit by a nurse, baby boys will be held with their legs hanging down, and baby girls will be held in hip flexion position.
  * Newborn with spontaneous voiding during the period from the beginning of the research procedure until the newborn is positioned will be excluded from the study.
  * The bladder stimulation technique will be repeated sequentially for 3 minutes until micturition begins.
  * After the maneuvers are started, the newborn's heart rate and saturation comfort scale score will be recorded at the 1st and 3rd minutes.
  * The success of the procedure and the duration of the procedure will be recorded
  Interventions: Procedure: The bladder stimulation technique
- Control Group (Active Comparator): * Newborns will be fed with formula or breast milk pumped, according to the age and weight of the baby.
  * Before the procedure, the newborn's heart rate, saturation and comfort scale score will be recorded.
  * Genital area will be cleaned.
  * Newborns will be fitted with a sterile urine bag suitable for their gender.
  * Babies who urinate spontaneously during the period until the sterile urine bag is fitted, the next feeding hour will be waited.
  * Newborn will be observed for 3 minutes. Newborn's heart rate and saturation comfort pain scale score will be recorded at the 1st and 3rd minutes.
  * The success of the procedure and the duration of the procedure will be recorded
  Interventions: Procedure: Steril urine bag

INTERVENTIONS:
Procedure: The bladder stimulation technique — The bladder stimulation technique consists of two consecutive maneuvers. In the first maneuver, the bladder is stimulated by tapping the suprapubic region for 30 seconds at a frequency of 100 touches per minute. In the second maneuver, circular massage is applied to the paravertebral region for 30 seconds. The two stimulation maneuvers will be repeated alternately for 3 minutes (180 seconds) until micturition begins. Maneuvers will be performed by the researcher. Infants in both groups will be held under the armpit by a parent, male infants will be held in the drooping legs, and female infants will be held in the hip flexion position.
  Arms: Experimental Group
Procedure: Steril urine bag — Steril urine bag are attached to the genital area to collect urine samples
  Other Names: Sterile urine bag
  Arms: Control Group

SUMMARY:
Urine specimen are necessary to diagnose various diseases in infants, especially urinary tract infections (UTI). Various non-invasive and invasive clinical interventions have been described for urine specimen collection. These; suprapubic aspiration, urinary catheterization, sterile urine collection bag and clean-caught urine (Herreros Fernández et al., 2013). For the diagnosis of UTI, it is recommended to collect urine samples by suprapubic aspiration (SPA) and urinary catheterization methods. However, these techniques are invasive and painful (Roberts et al. 2016). Clean-caught urine provides an acceptable urine sample for the diagnosis of UTI. But this method is possible for children with sphincter control. A technique was recently described that allows midstream urine specimen collection in children without sphincter control. This technique consists of bladder stimulation and lumbar paravertebral massage. The aim of this study is to evaluate the effect of bladder stimulation technique on procedural success, procedure time, physiological parameters and comfort in urine specimen collection in newborns.

DETAILED DESCRIPTION:
Urinary Tract Infection (UTI) is common in early childhood. Urinary Tract Infection (UTI) is the most common bacterial infection in febrile children younger than 3 months of age (Korbel et al., 2017; Velasco et al., 2015). A clean urine sample is required to diagnose various diseases, especially urinary tract infections (UTI) in infants. Various non-invasive and invasive clinical interventions have been described for urine specimen collection. These; suprapubic aspiration, urinary catheterization, sterile urine collection bag, and clean-caught urine (Herreros Fernández et al., 2013).

One of the non-invasive methods used to collect urine samples is the use of sterile urine collection bags (Herreros Fernández et al., 2013). This method is not an effective method due to its high false positive rate, time consuming, delayed treatment, skin irritation and high risk of contamination (Finnell et al., 2011; Kaufman et al., 2020). Therefore, sterile urine bags should be used in urinalysis instead of urine culture (Balighian & Review, 2018). Clean-caught urine provides an acceptable urine sample for the diagnosis of UTI. However, this method is possible for children with sphincter control (Altuntas et al., 2015; Kaufman et al., 2019).

A technique was recently described that allows midstream urine specimen collection in children without sphincter control. The technique, consisting of bladder stimulation and lumbar paravertebral massage, was successful in 86% of newborns, with an average duration of 57 seconds (Herreros Fernández et al., 2013). Previous studies have evaluated the technique's success rate and processing time (Altuntas et al., 2015, Labrosse et al., 2016, Crombie et al., 2020), contamination rate (Herreros et al., 2021), and cost (Kaufman et al., 2020) examined. Examination of the effect of the technique on the comfort and physiological parameters of the newborn will contribute to more information about the technique.

The aim of this study is to evaluate the effect of bladder stimulation technique on procedural success, procedure time, physiological parameters and comfort in urine specimen collection in newborns.

Study Population and Sampling The population of the research will be the newborns followed in the neonatal intensive care unit. The sample will consist of 64 (Experimental group = 32, Control group = 32) newborns who meet the inclusion criteria of the study. In calculating the sample size, Altuntaş et al. (2015) benefited from the study. Considering the success rates; The minimum number of samples to be taken was determined as 64 (Experimental group=32, Control group=32) with 95% confidence (1-α), 95% test power (1-β), w=0.453 effect size.

Randomization Infants meeting the research inclusion criteria will be divided into experimental and control groups using a computer-based program (https://www.randomizer.org).

Data Collection Method: The data will be collected by the a researcher in the unit where the study is planned to be carried out.

* Data Collection Form: Prepared by the researcher. The form includes questions about the infant's age, weight, gender, fever, heartbeat, saturation level, Comfortneo scale score, and procedure success and duration of the procedure.
* Comfortneo scale: Developed by Ambuel et al. (Ambuel et.al. 1992). Van Dijk et al. revised the COMFORTneo scale to measure behavior in newborns without physiological parameters (Van Dijk et. al. 2009). Turkish validity and reliability of the scale Kahraman et al. (Kahraman et. al 2014). The scale consists of 7 items: muscle tone, alertness, facial tension, calmness/agitation, body movements, respiratory response, and crying. "Respiratory response" is scored in infants on mechanical ventilator, and "crying" is scored in spontaneously breathing infants. A total score is calculated over 6 items. The lowest score that can be obtained from this scale is 6, and the highest score is 30. A high score indicates that the baby is not comfortable and needs interventions to provide comfort (Kahraman et. al 2014).
* Pulse Oximeter Device to detect infants' oxygen saturation (SPO2) and heart rate (HR)
* Weighing Tool to determine the current weight of babies.
* Thermometer to determine babies' body temperature

ELIGIBILITY:
Inclusion Criteria:

* Full-term newborns aged 3-28 days
* Collecting urine specimen
* Being fed orally
* Having written consent from parents

Exclusion Criteria:

* Poor general clinical condition (respiratory distress, etc.)
* Poor feding
* Dehydration
* Oliguria/anuria
* Treatment with nephrotoxic drugs
* Serious illnesses affecting the mobility of the baby
* Having neurological and anatomical anomalies that may affect bladder function Any condition (meningocele, meningomyelocele etc.) that will prevent the implementation of the stimulation maneuver

Ages: 3 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Procedural success | During the procedure (3 minutes)
  Procedural success is defined as urine sample collection within 3 minutes (180 seconds) of starting the stimulation maneuvers.
Duration of the procedure | During the procedure (3 minutes)
  Duration of the procedure is defined as the time from the beginning of bladder stimulation to the beginning of micturition

SECONDARY OUTCOMES:
Comfort | Before the procedure, at the 1st and 3rd minutes]
  The comfort levels of the newborns during the procedure will determined by the researcher.
Heart rate | Before the procedure, at the 1st and 3rd minutes]
  The heart rate of the infants will measured with hand portable pulse oximeter
Peripheral oxygen saturation level | Before the procedure, at the 1st and 3rd minutes]
  The peripheral oxygen saturation levels of the infants will measured with hand portable pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Narter Kaya, Principal Investigator — Kartal Dr. Lütfi Kirdar City Hospital; Birsen Mutlu, Principal Investigator — Istanbul University - Cerrahpasa; Nihan Korkmaz, Principal Investigator — Istanbul University - Cerrahpasa; Kadriye Şahin, Principal Investigator — Istanbul University - Cerrahpasa; Hande Özgürü, Principal Investigator — Kartal Dr. Lütfi Kirdar City Hospital
Locations (1):
- Nihan Korkmaz, Şişli, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Herreros Fernandez ML, Gonzalez Merino N, Tagarro Garcia A, Perez Seoane B, de la Serna Martinez M, Contreras Abad MT, Garcia-Pose A. A new technique for fast and safe collection of urine in newborns. Arch Dis Child. 2013 Jan;98(1):27-9. doi: 10.1136/archdischild-2012-301872. Epub 2012 Nov 21. PMID 23172785
- [Background] Korbel L, Howell M, Spencer JD. The clinical diagnosis and management of urinary tract infections in children and adolescents. Paediatr Int Child Health. 2017 Nov;37(4):273-279. doi: 10.1080/20469047.2017.1382046. Epub 2017 Oct 5. PMID 28978286
- [Background] Velasco R, Benito H, Mozun R, Trujillo JE, Merino PA, Mintegi S; Group for the Study of Febrile Infant of the RISeuP-SPERG Network. Febrile young infants with altered urinalysis at low risk for invasive bacterial infection. a Spanish Pediatric Emergency Research Network's Study. Pediatr Infect Dis J. 2015 Jan;34(1):17-21. doi: 10.1097/INF.0000000000000482. PMID 25036049
- [Background] SUBCOMMITTEE ON URINARY TRACT INFECTION. Reaffirmation of AAP Clinical Practice Guideline: The Diagnosis and Management of the Initial Urinary Tract Infection in Febrile Infants and Young Children 2-24 Months of Age. Pediatrics. 2016 Dec;138(6):e20163026. doi: 10.1542/peds.2016-3026. No abstract available. PMID 27940735
- [Background] Finnell SM, Carroll AE, Downs SM; Subcommittee on Urinary Tract Infection. Technical report-Diagnosis and management of an initial UTI in febrile infants and young children. Pediatrics. 2011 Sep;128(3):e749-70. doi: 10.1542/peds.2011-1332. Epub 2011 Aug 28. PMID 21873694
- [Background] Kaufman J. How to... collect urine samples from young children. Arch Dis Child Educ Pract Ed. 2020 Jun;105(3):164-171. doi: 10.1136/archdischild-2019-317237. Epub 2019 Aug 23. PMID 31444213
- [Background] Balighian E, Burke M. Urinary Tract Infections in Children. Pediatr Rev. 2018 Jan;39(1):3-12. doi: 10.1542/pir.2017-0007. No abstract available. PMID 29292282
- [Background] Altuntas N, Tayfur AC, Kocak M, Razi HC, Akkurt S. Midstream clean-catch urine collection in newborns: a randomized controlled study. Eur J Pediatr. 2015 May;174(5):577-82. doi: 10.1007/s00431-014-2434-z. Epub 2014 Oct 17. PMID 25319844
- [Background] Labrosse M, Levy A, Autmizguine J, Gravel J. Evaluation of a New Strategy for Clean-Catch Urine in Infants. Pediatrics. 2016 Sep;138(3):e20160573. doi: 10.1542/peds.2016-0573. Epub 2016 Aug 19. PMID 27542848
- [Background] Crombie T, Slinger R, Barrowman NJ, McGahern C, Smith L, Chu J, McCoy K, Akiki S, Agarwal A, Plint AC. Pragmatic evaluation of a midstream urine collection technique for infants in the emergency department. CJEM. 2020 Sep;22(5):665-672. doi: 10.1017/cem.2020.31. PMID 32383423
- [Background] Herreros ML, Gili P, Del Valle R, Barrios A, Pacheco M, Sanchez A. Urine collection methods for infants under 3 months of age in clinical practice. Pediatr Nephrol. 2021 Dec;36(12):3899-3904. doi: 10.1007/s00467-021-05142-4. Epub 2021 Jun 7. PMID 34100109
- [Background] Kaufman J, Knight AJ, Bryant PA, Babl FE, Dalziel K. Liquid gold: the cost-effectiveness of urine sample collection methods for young precontinent children. Arch Dis Child. 2020 Mar;105(3):253-259. doi: 10.1136/archdischild-2019-317561. Epub 2019 Aug 23. PMID 31444211
- [Background] Ambuel B, Hamlett KW, Marx CM, Blumer JL. Assessing distress in pediatric intensive care environments: the COMFORT scale. J Pediatr Psychol. 1992 Feb;17(1):95-109. doi: 10.1093/jpepsy/17.1.95. PMID 1545324
- [Background] van Dijk M, Roofthooft DW, Anand KJ, Guldemond F, de Graaf J, Simons S, de Jager Y, van Goudoever JB, Tibboel D. Taking up the challenge of measuring prolonged pain in (premature) neonates: the COMFORTneo scale seems promising. Clin J Pain. 2009 Sep;25(7):607-16. doi: 10.1097/AJP.0b013e3181a5b52a. PMID 19692803
- [Background] Kahraman A, Başbakkal Z, Yalaz M. Turkish Validity And Reliability Of Comfortneo Scale. International Refereed Journal of Nursing Research. 2014; 1: 1-11